CLINICAL TRIAL: NCT01876901
Title: Efficacy of Delayed Coloanal Anastomosis for Medium and Lower Rectum Cancer Treatment. Phase 2 Clinical Trial.
Brief Title: Efficacy of Delayed Coloanal Anastomosis for Medium and Lower Rectum Cancer Treatment. Phase 2 Clinical Trial (CASCADOR)
Acronym: CASCADOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB2010-08
Record Dates: First submitted 2012-11-05; First posted 2013-06-13 (Estimated); Results first posted 2021-08-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2021-07

CONDITIONS: Medium and Lower Rectal Cancer
Keywords: Rectal cancer; Coloanal anastomosis; Phase 2 clinical trial
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Two multicenter parallel single-arm phase II trials.
  One trial assessing 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA) in centers who routinely performing this intervention.
  One trial assessing colo-anal anastomosis (CAA) in centers who routinely performing this intervention.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA) (Experimental): Patients treated with 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA) in centers who routinely performing this intervention.
  Interventions: Procedure: 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA)
- Colo-anal anastomosis (CAA) (Experimental): Patients operated with colo-anal anastomosis (CAA) in centers who routinely performing this intervention.
  Interventions: Procedure: Colo-anal anastomosis (CAA)

INTERVENTIONS:
Procedure: 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA) — 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA) Whatever the mode of continuity restoration used, resection is the same in the two groups. It consists of total excision of the rectum and its mesorectum, that intervention should be performed by laparotomy or laparoscopy.
  After surgical resection, the colon is exteriorized through the anus and attached to the buttock.
  By day 6, exteriorized colon is resected and coloanal anastomosis is performed without preventive stoma derivation
  Arms: 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA)
Procedure: Colo-anal anastomosis (CAA) — After the surgical resection, coloanal anastomosis is performed usually after completion of a reservoir J when it is possible. Preventive ostomy is performed most often.
  In the absence of fistula, the patient will reoperation for stoma closure of its branch
  Arms: Colo-anal anastomosis (CAA)

SUMMARY:
Hypothesis:

In France, approximately 12,000 new rectal cancers are diagnosed each year. Frequency is one and a half times higher in men than in women. The average age of diagnosis is 65. Unlike colon cancer, technical management remains challenging with unresolved operating difficulties. Morbidity of surgical procedures remains high with a very large number of preventive or curative stoma derivations.

Reference in surgical treatment is total excision of the rectum and its mesentery, followed by continuity restoration by immediate coloanal anastomosis (ACAI). In this procedure, rate of fistula that results is reported in the literature between 15 and 25%.

An alternative to ACAI is delayed coloanal anastomosis without reservoir (ACAD). Based on retrospective experiences, we form the hypothesis that ACAD offers a much lower rate of fistula (<5%) and allows diminution of preventive stoma derivation practice. Morbidity and mortality are reduced, and patient's quality of life greatly improved. Direct costs (consumables intraoperative, hospitalization, stoma complications) and indirect (pocket-fitting stoma) are greatly reduced.

This study is a multicentre, two arms, phase 2 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven rectal adenocarcinoma.
* Medium or lower rectum tumour requiring removal of the entire rectum and its mesorectum.
* T1 N+ or T2 N+ or T3 N+ or T3 N0 and M0 tumour.
* Age between 18 and 75 years .
* ASA ≤ 2.
* Sphincter continence compatible with coloanal anastomosis.
* Patients who received preoperative radiotherapy alone or chemotherapy and radiotherapy.
* Patient affiliated to social security.
* For patients of childbearing age, use of contraception.
* Patient information and consent for study participation

Exclusion Criteria:

* Other histology of rectal cancer.
* T1 N0 or T2 N0 or T4 tumour.
* Metastatic disease M1.
* History of cancer except cervix in situ carcinoma or skin basal cell carcinoma.
* Patient with psychological, social, family or geographical reasons who couldn't be treated or monitored regularly by the criteria of the study
* Patients deprived of liberty or under guardianship.
* Pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-08-11 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: EVRARD Serge, PU-PH, Study Chair — Institut Bergonié
Locations (9):
- France (9):
  - CHU DE BORDEAUX - Hôpital Saint André, Bordeaux, Aquitaine
  - Institut Bergonié, Bordeaux, Aquitaine
  - CHU de GRENOBLE, Grenoble, Auvergne-Rhône-Alpes
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - HOSPICES CIVILS DE LYON - Hôpital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - Clinique Du Tonkin, Villeurbanne, Auvergne-Rhône-Alpes
  - Institut Paoli Calmettes, Marseille, Bouche Du Rhône
  - Chu de Nancy, Nancy, Lorraine
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy, Lorraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evrard S, Bellera C, Desolneux G, Cantarel C, Toulza E, Faucheron JL, Rivoire M, Dupre A, Mabrut JY, Bresler L, Marchal F, Bouriez D, Rullier E. Anastomotic leakage and functional outcomes following total mesorectal excision with delayed and immediate colo-anal anastomosis for rectal cancer: Two single-arm phase II trials. Eur J Surg Oncol. 2023 Nov;49(11):107015. doi: 10.1016/j.ejso.2023.107015. Epub 2023 Oct 23. PMID 37949519

RESULTS

PARTICIPANT FLOW:
Groups:
- 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA): Patients treated with 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA) in centers who routinely performing this intervention.
  2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA): 2-stage pull-through colo-anal anastomosis without prophylactic derivation (2SCA) Whatever the mode of continuity restoration used, resection is the same in the two groups. It consists of total excision of the rectum and its mesorectum, that intervention should be performed by laparotomy or laparoscopy.
  After surgical resection, the colon is exteriorized through the anus and attached to the buttock.
  By day 6, exteriorized colon is resected and coloanal anastomosis is performed without preventive stoma derivation
- Colo-anal Anastomosis (CAA): Patients operated with colo-anal anastomosis (CAA) in centers who routinely performing this intervention.
  Colo-anal anastomosis (CAA): After the surgical resection, coloanal anastomosis is performed usually after completion of a reservoir J when it is possible. Preventive ostomy is performed most often.
  In the absence of fistula, the patient will reoperation for stoma closure of its branch
Period: Overall Study
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Started | 65 | 59
Completed | 48 | 52
Not Completed | 17 | 7
Not completed — Protocol Violation | 10 | 2
Not completed — No or other surgical intervention | 7 | 5

BASELINE CHARACTERISTICS:
Population: Eligible patient (without major protocole deviation) which was operated with complete 2SCA procedure and CAA for 2SCA group and CAA group respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA) | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [56 to 67] | 63 [54 to 68] | 62 [55 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 29 | 28 | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 48 | 52 | 100

OUTCOME MEASURES:

1. Primary Outcome: Absence at Day 30 of a Symptomatic Anastomotic Leakage (AL) Among 2SCA
Description: Efficacy of the intervention was defined as the absence at day 30 of a symptomatic AL (either with entero-cutaneous fistula or perianastomotic abscess with infectious conditions and/or transit impairment) requiring diverting stoma (curatively for 2-stage CA or prophylactic-based for CA). AL was defined as fecal matter in the drainage system when a drainage system was present. Clinical signs included fever and subocclusion requiring a pelvic scan and collection of liquid and gas in the peri-anastomotic region. Non-symptomatic ALs which did not require any investigation nor treatment, in particular no diverting stoma, were not considered failures.
  Assuming an efficacy rates of 85% (null hypothesis) and 95% (alternative hypothesis), and relied on a superiority test at the 5% significance level (one-sided) with 80% power, 53 eligible and assessable patients were required. Efficacy of the intervention was concluded if at least 49 patients had no symptomatic AL at day 30.
Time Frame: Delayed coloanal anastomosis effectiveness was evaluated in terms of symptomatic anastomotic fistula occurring during the 30 days post anastomosis and requiring stoma derivation.
Population: Eligible patient (without major protocol deviation) which was operated with complete 2SCA procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA)
Number analyzed (Participants) | 48
Participants | 1

2. Secondary Outcome: Stomata Bypass (Preventive or Therapeutic)
Description: Number of patients with stomata bypass (preventive or therapeutic) at each time of follow-up after surgery (2SCA or CAA).
  A stomata bypass is the result of a surgical operation in which a damaged part is removed from the ileum (ileostomy) or colon (colostomy) and the cut end diverted to an artificial opening in the abdominal wall.
Time Frame: Presence of stomata bypass was evaluated at 30 days, 1 year and 2 years after surgery (2SCA or CAA)
Population: Eligible patient (without major protocol deviation) which was operated with complete 2SCA procedure and CAA for 2SCA group and CAA group respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 48 | 52
Participants
  30 days | 2 | 49
  1 year | 3 | 3
  2 years | 6 | 8

3. Secondary Outcome: Post-operative Morbidity
Description: Post-operative morbidity was assessed in terms number of patients with at least one surgical complications related to treatment and related to a serious adverse event.
Time Frame: During the 30 first days after surgery (2SCA or CAA)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 48 | 52
Participants | 13 | 10

4. Secondary Outcome: Postoperative Mortality
Description: Postoperative mortality was defined by the number of patients who deceased (all cause mortality) during the first 30 days after surgery (2SCA or CAA).
Time Frame: From the date of surgery to 30 days after surgery (2SCA or CAA)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 48 | 52
Participants | 0 | 0

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the date of surgery and the date of the earliest of the following events:
  * The patient's death, whatever the cause,
  * Local progression or remotely.
  Progression was defined as clinical or radioglogical progression. Radiological progression was defined Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions"
  1-year and 2-year progression-free rates were estimated.
Time Frame: 1 and 2 years after surgery (2SCA or CAA)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage or paticipants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 48 | 52
percentage or paticipants
  1-year PFS | 76.5 [61.5 to 86.2] | 92.2 [80.6 to 97.0]
  2-years PFS | 63.3 [47.7 to 75.4] | 81.3 [66.9 to 89.9]

6. Secondary Outcome: Number of Participants With Anal Incontinence at 6 Months
Description: The digestive functions, especially anal incontinence was evaluated according to the scale of 5 items Jorge and Wexner (score from 0 to 20).
  The rate of patients with anal incontinence (score >=5) at 6 months was reported.
Time Frame: At 6 months after surgery (2SCA or CAA)
Population: Eligible patient (without major protocol deviation) which was operated with complete 2SCA procedure and CAA for 2SCA group and CAA group respectively and who responded to the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 25 | 39
Participants | 25 | 32

7. Secondary Outcome: Number of Participants With Anal Incontinence at 12 Months
Description: The digestive functions, especially anal incontinence was evaluated according to the scale of 5 items Jorge and Wexner (score from 0 to 20).
  The rate of patients with anal incontinence (score >=5) at 12 months was reported.
Time Frame: At 12 months after surgery (2SCA or CAA)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 16 | 40
Participants | 15 | 36

8. Secondary Outcome: Number of Participants With Anal Incontinence at 24 Months
Description: The digestive functions, especially anal incontinence was evaluated according to the scale of 5 items Jorge and Wexner (score from 0 to 20).
  The rate of patients with anal incontinence (score >=5) at 24 months was reported.
Time Frame: At 24 months after surgery (2SCA or CAA)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 12 | 33
Participants | 11 | 29

9. Secondary Outcome: Absence at Day 30 of a Symptomatic Anastomotic Leakage (AL) Among CAA
Description: Efficacy of the intervention was defined as the absence at day 30 of a symptomatic AL (either with entero-cutaneous fistula or perianastomotic abscess with infectious conditions and/or transit impairment) requiring diverting stoma. AL was defined as fecal matter in the drainage system when a drainage system was present. Clinical signs included fever and subocclusion requiring a pelvic scan and collection of liquid and gas in the peri-anastomotic region. Non-symptomatic ALs which did not require any investigation nor treatment, in particular no diverting stoma, were not considered failures.
  The effectiveness of the CAA surgery will be evaluated in terms of absence of fistula requiring stoma diversion. Similarly to 2SCA group, 53 CAA eligible and evaluable patients will be required. If 49 or more patients (out of 53) have no fistula requiring stoma diversion, then we conclude that the CAA is effective. To anticipate any non evaluable patients, we plan to recruit 58 patients CAA.
Time Frame: Colo-anal anastomosis effectiveness will be evaluated in terms of symptomatic anastomotic fistula occurring during the 30 days post anastomosis and requiring stoma derivation.
Population: Eligible patient (without major protocol deviation) which was operated with complete CAA procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Colo-anal Anastomosis (CAA)
Number analyzed (Participants) | 52
Participants | 5

ADVERSE EVENTS:
Time Frame: From dated written informed consents, up to 30 days following last follow-up, with an average of 24 months.
Description: Only Serious Adverse events were collected following NCI-CTCAE (3.0).
  Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) | Colo-anal Anastomosis (CAA)
All-Cause Mortality (participants affected / at risk) | 4/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 30/48 | 24/52
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-stage Pull-through Colo-anal Anastomosis Without Prophylactic Derivation (2SCA) (N=48) | Colo-anal Anastomosis (CAA) (N=52)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0) — CARDIAC GENERAL
ALTERED GENERAL CONDITION (General disorders) | 2 (2) | 1 (1) — CONSTITUTIONAL SYMPTOMS
ABDOMINO PERINEAL AMPUTATION FOR RECURRENCE OF RECTAL ADENOCARCINOMA (Surgical and medical procedures) | 1 (1) | 0 (0) — CONSTITUTIONAL SYMPTOMS
MANAGEMENT OF HEPATIC METASTASES OF THE ANTERIOR BORDER OF SEGMENT VII (Surgical and medical procedures) | 1 (1) | 0 (0) — CONSTITUTIONAL SYMPTOMS
LEFT COLON LUMPECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) — CONSTITUTIONAL SYMPTOMS
Hepatic metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — CONSTITUTIONAL SYMPTOMS
DISEASE PROGRESSION (General disorders) | 0 (0) | 0 (0) — CONSTITUTIONAL SYMPTOMS
METACHRONOUS LIVER METASTASES OF RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — CONSTITUTIONAL SYMPTOMS
Metastatic recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — CONSTITUTIONAL SYMPTOMS
ANASTOMOTIC RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — CONSTITUTIONAL SYMPTOMS
LOCAL AND METASTATIC RECURRENCE (LUNGS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — CONSTITUTIONAL SYMPTOMS
HEPATIC EVOLUTIONARY RECOVERY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — CONSTITUTIONAL SYMPTOMS
PELVIC TUMOR RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — CONSTITUTIONAL SYMPTOMS
PERISTOMAL DERMATITIS ASSOCIATED WITH SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — DERMATOLOGY/SKIN
Ascites (non-malignant) (Gastrointestinal disorders) | 0 (0) | 1 (1) — GASTROINTESTINAL
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — GASTROINTESTINAL
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — GASTROINTESTINAL
Fistula, GI (Gastrointestinal disorders) | 2 (2) | 4 (5) — GASTROINTESTINAL
Anitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — GASTROINTESTINAL
RECTAL RESECTION SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1) — GASTROINTESTINAL
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 0 (0) | 2 (2) — GASTROINTESTINAL
Incontinence, anal (Gastrointestinal disorders) | 0 (0) | 3 (3) — GASTROINTESTINAL
Necrosis, GI (Gastrointestinal disorders) | 2 (2) | 0 (0) — GASTROINTESTINAL
Obstruction, GI (Gastrointestinal disorders) | 6 (6) | 3 (3) — GASTROINTESTINAL
Stricture/stenosis (including anastomotic), GI (Gastrointestinal disorders) | 4 (4) | 3 (4) — GASTROINTESTINAL
Hematoma (Vascular disorders) | 2 (3) | 1 (1) — HEMORRHAGE/BLEEDING
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — HEMORRHAGE/BLEEDING
Infection with unknown ANC (Infections and infestations) | 13 (20) | 12 (18) — INFECTION
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0) — NEUROLOGY
Cognitive disturbance (Psychiatric disorders) | 0 (0) | 1 (1) — NEUROLOGY
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 (1) | 0 (0) — NEUROLOGY
Pain (General disorders) | 1 (1) | 0 (0) — PAIN
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — PULMONARY/UPPER RESPIRATORY
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — PULMONARY/UPPER RESPIRATORY
Stricture/stenosis (including anastomotic), GU (Renal and urinary disorders) | 1 (1) | 0 (0) — RENAL/GENITOURINARY
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2) | 2 (2) — RENAL/GENITOURINARY
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2) — SEXUAL/REPRODUCTIVE FUNCTION
EVENTRATION (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) — SURGERY/INTRA-OPERATIVE INJURY
BILATERAL INGUINAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — SURGERY/INTRA-OPERATIVE INJURY
STOMAL PROLAPSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — SURGERY/INTRA-OPERATIVE INJURY
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) — VASCULAR
Visceral arterial ischemia (non-myocardial) (Vascular disorders) | 1 (1) | 2 (2) — VASCULAR

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT01876901/Prot_SAP_000.pdf